CLINICAL TRIAL: NCT06867341
Title: Monocentric Prospectiv Observational Clinical Trial of Pelvic Floor Biometry During Pregnancy and Puerperium : Relationship with Symptoms Related to Post-partum Pelvic Floor Dysfunction
Brief Title: Monocentric Prospectiv Observational Clinical Trial of Pelvic Floor Biometry During Pregnancy and Puerperium
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Arsenio Spinillo, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PavPel
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Disorders; Pelvic Floor Distress and Impact Scores
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PREGNAANT WOMEN

SUMMARY:
Pregnancy, childbirth and the puerperium determine significant changes in the muscular, fascial and support structures of the pelvic floor. These changes, both physiological (i.e. dictated by the adaptations that pregnancy determines at the level of the connective tissue, collagen and pelvic-perineal muscular structures) and the changes induced by the passage of the fetus through the birth canal (obstetric lacerations, episiotomy and muscle avulsions) cause a weakening of the pelvic support structures with the possible onset of dysfunctional symptoms, which are not only common in old age, but become evident already in childbearing age. Previous studies on the composition of connective tissue show significant changes in the collagen component both in continent women and in those who experience stress urinary incontinence. These changes are revealed in approximately 24% of the population that suffers from urinary incontinence. Collagen is the main component of the endopelvic fascia. During pregnancy, the hormonal influence typical of this phase determines significant changes in the mechanical properties of the connective tissue and muscle fibers of the levator ani, which tend to hypertrophy and lengthen. This may also explain why cesarean delivery, elective or after the onset of labor, is not fully protective against the development of pelvic floor dysfunction. However, pelvic floor changes may have occurred before delivery and may not necessarily be related to labor and delivery itself. Incontinence, mostly temporary in pregnancy, must be interpreted as the result of these factors in addition to the increased pressure on the urethrovesical junction caused by the gravid uterus. Stretching of connective tissues beyond their physiological limits during labor, resulting in levator ani injury and/or possible neurogenic stretch damage, occurs in the majority of women who give birth vaginally, but in most women, muscle hypertrophy and nerve fiber adaptation compensate for this pathological pattern. In a minority (5-20%) of women, major levator ani defects and neurogenic lesion may lead to irreversible changes in pelvic floor function. Pelvic floor imaging after pregnancy has improved the understanding of the etiology of pelvic floor disorders in animal models. Patients who already present with pelvic static dysfunction and urinary incontinence during pregnancy tend to develop the same problems in the puerperium. However, to date it is not known what moment in pregnancy these changes in the pelvic tissue begin and that cause the progressive change in the myo-connective components of pregnancy. The lack of prospective cohort studies of pregnant and postpartum subjects does not allow a conclusive opinion on this topic. Pelvic floor ultrasound performed transpeineally, useful for evaluating pelvic biometry, is a non-invasive method and well tolerated by the patient, not only in postpartum but also during pregnancy. A previous study examined pelvic floor changes during pregnancy, reporting how the progression of pregnancy determines changes in the anatomical components of the pelvic floor, without however correlating the data with the puerperium and the longer-term outcomes of these changes. We did not identify any previously published studies that attempted to comprehensively assess biometric changes of the pelvic floor during pregnancy and postpartum using not only ultrasound imaging, but also clinical assessment and validated urinary symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy confirmed by ultrasound in the first trimester (within 10 weeks of gestational age),
* maternal age between 18 and 40 years,
* patients who speak Italian correctly and/or who can perfectly understand what was expressed at the time of enrollment.
* spontaneous vaginal births, operative and current cesarean section
* patients who do not report urinary and fecal incontinence or pelvic organ prolapse at enrollment.

Exclusion Criteria:

* previous pregnancy ended with spontaneous vaginal delivery or cesarean section
* pelvic floor reconstructive surgery
* gynecological cancer
* pelvic radiation therapy for previous oncological disease
* previous pelvic trauma
* known connective tissue disease
* body mass index >40 kg / m2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be consecutively enrolled in the three trimesters of pregnancy and in the puerperium, nulliparous, and who did not report pelvic static disorders at the time of enrollment (fecal and urinary incontinence and symptoms of genital prolapse).
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
pelvic floor biometry | baseline, at second trimester of pregnancy, at third trimester of pregnancy, six weeks after delivery
  evaluate the association between the biometry of the pelvic floor and the presence of symptoms such as urinary and fecal incontience, pelvic weight and vaginal congestion typical of genital prolapse, related to pelvic-perineal dysfunction at the check-up carried out 6 months after delivery. Specifically, the following end-points will be evaluated: pelvic hiatus area, measured in the last trimester of pregnancy and in the post-partum

SECONDARY OUTCOMES:
pelvic floor biometry | baseline, at second trimester of pregnancy, at third trimester of pregnancy, six weeks after delivery
  1. time course of the pelvic hiatus area
  2. time course of the anteroposterior diameter
  3. time course of the transverse diameter of the pelvic hiatus
  4. time course of the presence/intensity of symptoms based on the score obtained in the PDFI questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Ostetricia e Ginecologia 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Solans-Domenech M, Sanchez E, Espuna-Pons M; Pelvic Floor Research Group (Grup de Recerca del Sol Pelvia; GRESP). Urinary and anal incontinence during pregnancy and postpartum: incidence, severity, and risk factors. Obstet Gynecol. 2010 Mar;115(3):618-628. doi: 10.1097/AOG.0b013e3181d04dff. PMID 20177295
- [Background] Costantini S, Esposito F, Nadalini C, Lijoi D, Morano S, Lantieri P, Mistrangelo E. Ultrasound imaging of the female perineum: the effect of vaginal delivery on pelvic floor dynamics. Ultrasound Obstet Gynecol. 2006 Feb;27(2):183-7. doi: 10.1002/uog.2663. PMID 16388512